CLINICAL TRIAL: NCT01164891
Title: A Phase I, Open-label, Excretion Balance, Pharmacokinetic and Metabolism Study After Single Oral Dose of 14C-labeled RO5185426 in Previously Treated and Untreated Patients With Metastatic Melanoma
Brief Title: A Pharmacokinetic and Metabolism Study of 14C-labeled RO5185426 on Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25158
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5185426

INTERVENTIONS:
Drug: RO5185426 — Continuous oral dosing b.i.d. , on Day 15 a C isotope labeled dose will be administered

SUMMARY:
This open-label, non-randomized study will assess the mass balance, metabolism, routes and rates of elimination as well as efficacy and safety of RO5185426 (RG7204; PLEXXIKON; PLX4032) in previously treated or untreated patients with metastatic melanoma. Patients will receive continuous twice daily oral treatment with RO5185426. On Day 15, a 14C-labeled dose will be administered. Anticipated time on study treatment is until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed metastatic melanoma, surgically incurable and unresectable Stage IIIc or IV (AJCC)
* Prior treatment for metastatic melanoma allowed; >/= 28 days must be elapsed since previous systemic treatment prior to first administration of study drug
* Positive BRAF V600E mutation result (by Roche CoDx test)
* ECOG performance status 0-1
* Adequate hematologic, renal and liver function
* Body Mass Index (BMI) 18 to 32 kg/m2 inclusive

Exclusion Criteria:

* Active CNS lesions
* History of or known spinal cord compression, or carcinomatous meningitis
* Anticipated or ongoing administration of any anticancer therapies other than those administered in this study
* Refractory nausea or vomiting, or other medical conditions that are capable of altering the absorption, metabolism or elimination of the study drug
* Known clinically significant active infection
* Known HIV positivity or AIDS-related illness, active HBV, or active HCV
* Previous malignancy within the past 5 years, except for basal or squamous cell carcinoma of the skin, melanoma in situ, and carcinoma in situ of the cervix
* Clinically significant cardiovascular disease or incident within the 6 months prior to study drug administration
* Patients who have had at least one dose of study drug (RO5185426 or comparator) in a clinical trial that includes RO5185426

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- 14C-labeled RO5185426: Participants received non-labeled RO5185426 film-coated tablets 960 milligrams (mg) orally two times daily (BID) from Day 1 to Day 14. On Day 15, participants received a single dose of 960 mg RO5185426 with a maximum of 2.56 millibecquerel (69.2 microcurie) of 14C RO5185426. After Day 15, participants received non-labeled RO5185426 film-coated tablets 960 mg orally BID until the development of progressive disease, unacceptable toxicity, consent withdrawal, death, lost to follow-up or any other criteria for removal as determined by the investigator.
Period: Overall Study
Arm/Group | 14C-labeled RO5185426
Started | 7
Completed | 1
Not Completed | 6
Not completed — Disease Progression | 5
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants were analyzed.
Groups:
- 14C-labeled RO5185426: Participants received non-labeled RO5185426 film-coated tablets 960 mg orally BID from Day 1 to Day 14. On Day 15, participants received a single dose of 960 mg RO5185426 with a maximum of 2.56 millibecquerel (69.2 microcurie) of 14C RO5185426. After Day 15, participants received non-labeled RO5185426 film-coated tablets 960 mg orally BID until the development of progressive disease, unacceptable toxicity, consent withdrawal, death, lost to follow-up or any other criteria for removal as determined by the investigator.
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma RO5185426 Trough Concentrations on Days 15,16, and 17
Time Frame: Pre-dose on Days 15, 16 and 17
Population: Pharmacokinetic (PK) Analysis Population: participants from whom the level of radioactivity recovered from excreta (urine and feces) was ≤ 1% of the radioactivity in the administered dose between any two successive 48-hour interval assessments.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
micrograms per milliliter
  Day 15 | 61.1 (28.1)
  Day 16 | 67.7 (22.2)
  Day 17 | 61.5 (13.4)

2. Secondary Outcome: Number of Participants With a Response by Confirmed Best Overall Response
Description: Best overall response (according to Response Evaluation Criteria In Solid Tumors 1.1 criteria) was defined as best response recorded from start of treatment until disease progression which included complete response (CR) or partial response (PR) that had been confirmed by second tumor assessment no less than (<) 4 weeks after criteria for response were first met. Confirmed CR: disappearance of all target and non-target lesions; no new lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeters (mm). Confirmed PR: at least 30% decrease in sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Disease progression: at least 20% increase in sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: From Baseline then Day 1 of Cycle 3 thereafter, Day 1 of every other cycle (every 2 months) until disease progression, withdrawal from study or death (maximum 841 days)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
participants | 4

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of first treatment to the date of death, regardless of the cause of death.
Time Frame: From Baseline then Day 1 of Cycle 3 thereafter, Day 1 of every other cycle (every 2 months) until death (maximum 841 days)
Population: The data was not collected, as planned, due to small number of participants enrolled in the study.
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 0

4. Primary Outcome: Maximum Plasma Concentration of 14C-labeled RO5185426 (Cmax) in Both Blood and Plasma
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). 14C-labeled RO5185426 given was equivalent to ≤1 millisieverts (mSv).
Time Frame: 0 hour (prior to evening dose) on Day 14; 0 hour (pre dose), 1, 2, 4, 6, 12, 24, 36, 48, 72, 96, 168, 216, 312 hours post dose on Day 15, and then every 96 hour until recovery criteria met (maximum: 432 hours)
Population: PK Analysis Population. Number of participants analyzed = participants with measurable data for this outcome.
Measure: Mean (Standard Deviation); unit: micrograms equivalent per milliliter
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 5
micrograms equivalent per milliliter
  Blood | 5.25 (1.71)
  Plasma | 7.83 (2.28)

5. Primary Outcome: Time to Reach Cmax in Both Blood and Plasma
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments).
Time Frame: as for outcome 4
Population: PK Analysis Population. Number of participants analyzed = participants with measurable data for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 5
hours
  Blood | 4.1 [4.0 to 12.0]
  Plasma | 4.1 [4.0 to 12.0]

6. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Sample (AUClast) of 14C-RO5185426 in Both Blood and Plasma
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). 14C-labeled RO5185426 given was equivalent to ≤1mSv.
Time Frame: as for outcome 4
Population: PK Analysis Population. Number of participants analyzed = participants with measurable data for this outcome.
Measure: Mean (Standard Deviation); unit: (micrograms equivalent/milliliter)*hour
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 5
(micrograms equivalent/milliliter)*hour
  Blood | 456.0 (85.4)
  Plasma | 633.0 (123.0)

7. Primary Outcome: Half-life of 14C-labeled RO5185426 in Both Blood and Plasma
Description: as for outcome 5
Time Frame: as for outcome 4
Population: PK Analysis Population. Number of participants analyzed = participants with measurable data for this outcome.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 5
hour
  Blood | 84.4 (24.6)
  Plasma | 71.1 (15.4)

8. Primary Outcome: AUC Ratio of Blood:Plasma 14C-labeled RO5185426
Description: as for outcome 5
Time Frame: as for outcome 4
Population: PK Analysis Population. Number of participants analysed = participants with measurable data for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 5
ratio | 0.72 (0.05)

9. Primary Outcome: 14C-labeled RO5185426 Recovery: Percentage of Dose Excreted in Feces and Urine
Description: Urinary and fecal samples were analyze for the percentage dose recovered as total radioactivity. The radioactivity was determined on a Packard liquid scintillation counter. Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments).
Time Frame: Urine:0 hour (pre dose),in quantitative fraction(0-6,6-12,12-24 hours) post dose on Day 15,during 24 hour interval thereafter;Feces:From Day 14 upto pre dose on Day 15,during 24 hour interval post dose until recovery criterion;(maximum:432 hours for both)
Population: PK Analysis Population. One participant was excluded in the analysis because of contamination of urine sample with feces.
Measure: Mean (Standard Deviation); unit: percentage of dose recovered
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 6
percentage of dose recovered
  Percent Dose Recovery in Feces | 94.05 (2.66)
  Percent Dose Recovery in Urine | 0.97 (0.43)
  Percent Dose Total Recovery (Feces and Urine) | 95.02 (2.40)

10. Primary Outcome: Percentage of Total Integrated Radioactivity in Plasma of 14C-labeled RO5185426 and 14C-labeled Metabolite
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). Plasma samples were pooled over three time intervals for this analysis based on available radioactive counts (4 + 6 hours, 12 + 24 hours, and 36 + 48 hours). Radioactivity was measured in terms of region of interest by high performance liquid chromatography. The radiolabelled components in each chromatogram were evaluated to determine retention times and peak area values. Data for 14C-labeled RO5185426 and 14C-labeled metabolite (mono-hydroxy) are reported.
Time Frame: 4+6 hours, 12 +24 hours, 36+48 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
percentage of total radioactivity
  RO5185426: 4 + 6 hours | 99.46 (1.42)
  RO5185426: 12 + 24 hours | 95.93 (5.49)
  RO5185426: 36 + 48 hours | 96.03 (3.76)
  Mono-hydroxy Metabolite: 4 + 6 hours | 0.54 (1.42)
  Mono-hydroxy Metabolite: 12 + 24 hours | 4.07 (5.49)
  Mono-hydroxy Metabolite: 36 + 48 hours | 3.97 (3.76)

11. Primary Outcome: Plasma 14C-labeled RO5185426 and 14C-labeled Metabolite Levels
Description: Collection of samples for radioactivity continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48 hour interval assessments). Plasma samples were pooled over three time intervals for this analysis based on available radioactive counts (4 + 6 hours, 12 + 24 hours, and 36 + 48 hours). The concentrations were measured in nanogram equivalent per gram which was calculated based on ratio of dosed radioactivity and the last dose of RO5185426. The concentration values represented the drug portion of the last dose. Data for 14C-labeled RO5185426 and 14C-labeled metabolite (mono-hydroxy) are reported.
Time Frame: 4+6 hours, 12 +24 hours, 36+48 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: nanogram equivalent per gram
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
nanogram equivalent per gram
  RO5185426: 4 + 6 hours | 6122 (2537)
  RO5185426: 12 + 24 hours | 6139 (1787)
  RO5185426: 36 + 48 hours | 4710 (1544)
  Mono-hydroxy Metabolite: 4 + 6 hours | 57 (152)
  Mono-hydroxy Metabolite: 12 + 24 hours | 321 (442)
  Mono-hydroxy Metabolite: 36 + 48 hours | 238 (249)

12. Primary Outcome: Percentage of Total Integrated Radioactivity in Feces of 14C-labeled RO5185426 and 14C-labeled Metabolite
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). Fecal samples were pooled over two time intervals for this analysis (0-24 + 24-48 hours, 48-72 + 72-96 hours). Radioactivity was measured in terms of region of interest by high performance liquid chromatography. The radiolabelled components in each chromatogram were evaluated to determine retention times and peak area values. Data for 14C-labeled RO5185426 and 14C-labeled metabolites (glucosylation, mono-hydroxy, and glucuronide) are reported.
Time Frame: 0-24 + 24-48 hours, 48-72 + 72-96 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Groups:
- 14C-labeled RO5185426: Participants received non-labeled RO5185426 film-coated tablets 960 mg orally BID from Day 1 to Day 14. On Day 15 participants received a single dose of 960 mg RO5185426 with a maximum of 2.56 millibecquerel (69.2 microcurie) of 14C RO5185426. After Day 15, participants received non-labeled RO5185426 film-coated tablets 960 mg orally BID until the development of progressive disease, unacceptable toxicity, consent withdrawal, death, lost to follow-up or any other criteria for removal as determined by the investigator.
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
percentage of total radioactivity
  RO5185426: 0-24 + 24-48 hours | 94.19 (5.75)
  RO5185426: 48-72 + 72-96 hours | 55.52 (20.12)
  Glucosylation: 0-24 + 24-48 hours | 2.58 (3.06)
  Glucosylation: 48-72 + 72-96 hours | 18.83 (6.71)
  Mono-hydroxy: 0-24 + 24-48 hours | 0.15 (0.41)
  Mono-hydroxy: 48-72 + 72-96 hours | 13.71 (9.07)
  Glucuronide: 0-24 + 24-48 hours | 3.08 (4.01)
  Glucuronide: 48-72 + 72-96 hours | 11.94 (12.13)

13. Primary Outcome: Percentage of Total Dose in 14C-labeled RO5185426 and 14C-labeled Metabolite in Pooled Fecal Samples
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). Fecal samples were pooled over 2 time intervals (0-24 + 24-48 hours, 48-72 + 72-96 hours) for measurement of 14C-labeled RO5185426 and 14C-labeled metabolites (glucosylation, mono-hydroxy, glucuronide) levels.
Time Frame: 0-24 + 24-48 hours, 48-72 + 72-96 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: percentage of total dose administered
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
percentage of total dose administered
  RO5185426: 0-24 + 24-48 hours | 37.49 (21.59)
  RO5185426: 48-72 + 72-96 hours | 17.10 (11.45)
  Glucosylation: 0-24 + 24-48 hours | 0.97 (1.08)
  Glucosylation: 48-72 + 72-96 hours | 5.04 (2.91)
  Mono-hydroxy: 0-24 + 24-48 hours | 0.11 (0.29)
  Mono-hydroxy: 48-72 + 72-96 hours | 3.30 (2.23)
  Glucuronide: 0-24 + 24-48 hours | 1.19 (1.42)
  Glucuronide: 48-72 + 72-96 hours | 2.86 (3.13)

14. Primary Outcome: Percentage of Total Integrated Radioactivity in Urine of 14C-labeled RO5185426 and 14C-labeled Metabolite
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). Urine samples were pooled over period of 96 hours (pool of 0-6 + 6-12 + 12-24 + 24-48 + 48-72 + 72-96 hour samples), Radioactivity was measured in terms of region of interest by high performance liquid chromatography. The radiolabelled components in each chromatogram were evaluated to determine retention times and peak area values. Data for 14C-labeled RO5185426 and 14C-labeled metabolites (2 unknown metabolites, glucosylation, mono-hydroxy) are reported.
Time Frame: 0 up to 96 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
percentage of total radioactivity
  RO5185426 | 32.38 (37.30)
  Unknown Metabolite 1 | 4.56 (12.05)
  Unknown Metabolite 2 | 25.44 (35.51)
  Glucosylation | 30.22 (28.79)
  Mono-hydroxy | 7.41 (12.87)

15. Primary Outcome: Percentage of Total Dose in 14C-labeled RO5185426 and 14C-labeled Metabolite in Pooled Urine Samples
Description: Collection of samples continued until the recovery criterion was met (radioactivity recovered from urine and feces ≤ 1 % of the radioactivity in the administered dose between any two successive 48-hour interval assessments). Urine samples were pooled over period of 96 hours (pool of 0-6 + 6-12 + 12-24 + 24-48 + 48-72 + 72-96 hour samples). Data for parent drug (RO5185426) and metabolites (2 unknown metabolites, glucosylation, mono-hydroxy) are reported.
Time Frame: 0 up to 96 hours post dose on Day 15
Population: PK Analysis Population.
Measure: Mean (Standard Deviation); unit: percentage of total dose administered
Arm/Group | 14C-labeled RO5185426
Number analyzed (Participants) | 7
percentage of total dose administered
  RO5185426 | 1.03 (2.33)
  Unknown Metabolite 1 | 0.04 (0.10)
  Unknown Metabolite 2 | 0.17 (0.21)
  Glucosylation | 0.24 (0.26)
  Mono-hydroxy | 0.05 (0.10)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose (up to 869 days)
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | 14C-labeled RO5185426
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 14C-labeled RO5185426 (N=7)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 14C-labeled RO5185426 (N=7)
Anemia (Blood and lymphatic system disorders) | 1
Conjunctivital Hyperaemia (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Lip Swelling (Gastrointestinal disorders) | 1
Parotid Gland Enlargement (Gastrointestinal disorders) | 1
Tongue Coated (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Device Related Infection (Infections and infestations) | 1
Erythema Induratum (Infections and infestations) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Blood Potassium Decreased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Weight Decreased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Follicular (Skin and subcutaneous tissue disorders) | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.